CLINICAL TRIAL: NCT01146171
Title: A Phase I Multiple Ascending Dose Study of BMS-844203 (CT-322) Monotherapy in Japanese Patients With Solid Tumors
Brief Title: Japanese Phase 1 Study of BMS-844203 (CT322)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA196-007
Record Dates: First submitted 2010-06-10; First posted 2010-06-17 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — CT-322

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-844203 (CT-322) (Experimental)
  Interventions: Drug: BMS-844203 (CT-322)

INTERVENTIONS:
Drug: BMS-844203 (CT-322) — Injection, IV, 1 and 2 mg/kg, Weekly, Until disease progression or unacceptable toxicity became apparent

SUMMARY:
The purpose of this clinical study is to evaluate the safety and tolerability of CT-322 monotherapy to determine the recommended dose for phase II and subsequent studies

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid tumors for whom the standard of care is ineffective or inappropriate
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group performance 0-1

Exclusion Criteria:

* Subject has uncontrolled diabetes or hypertension
* Clinical significant bleeding diathesis or coagulopathy
* Thrombotic or embolic cerebrovascular accident

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Determine recommended dose for Phase 2 study of CT-322 | Within the first 28 days

SECONDARY OUTCOMES:
To assess the plasma pharmacokinetics of CT-322. Pharmacokinetics of CT-322 will be derived from plasma concentration versus time data. The pharmacokinetic parameters to be assessed include Cmax, Cmin, Tmax, AUC (INF), AUC (TAU), T-HALF, etc. | Cycle 1: Day 1 to 5, 8, 15, 22 to 26 and 29
To assess the plasma pharmacokinetics of CT-322. Pharmacokinetics of CT-322 will be derived from plasma concentration versus time data. The pharmacokinetic parameters to be assessed include Cmax, Cmin, Tmax, AUC (INF), AUC (TAU), T-HALF, etc. | Cycle 2 and beyond (up to 6 cycle): Day 1 at each cycle and then every 3 cycles thereafter
To assess anti-tumor activity of CT-322 | Every 8 weeks
To assess the effects of CT-322 on plasma VEGF levels | Cycle 1: Day 1, 3, 8, 15, 22
To assess the effects of CT-322 on plasma VEGF levels | Cycle 3: Day 1
To assess the presence of anti CT-322 antibodies | Cycle 1: Day 1, 15, 22 and 29
To assess the presence of anti CT-322 antibodies | Cycle 3 and beyond (up to 6 cycle): Day 1 at each cycle and then every 3 cycles thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Osaka-Sayama-Shi, Osaka, Japan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx